CLINICAL TRIAL: NCT00265681
Title: Proactive Telephone Counseling With Rural Smokeless Tobacco Users
Brief Title: Telephone Counseling for Snuff Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Minnesota Partnership for Action Against Tobacco (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-119; RC -2004-0010
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2007-04

CONDITIONS: Smokeless Tobacco; Tobacco Use Cessation
Keywords: smokeless tobacco cessation; chewing tobacco; oral tobacco; smokeless tobacco; telephone; counseling
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Phone counseling and written materials

SUMMARY:
The primary objective is to evaluate the effectiveness of telephone-based counseling in promoting smokeless tobacco cessation among residents of Minnesota. It is hypothesized that a greater proportion of individuals assigned to the proactive telephone calls will quit their use of smokeless tobacco products and all tobacco products compared to the comparison group not receiving those calls.

DETAILED DESCRIPTION:
Smokeless Tobacco (ST) users have not been the focus of tobacco control campaigns in Minnesota. However, there are a significant number of adults in Minnesota who regularly use ST. There is a need for a low-cost cessation program that can be widely delivered to ST users who may have little or no access to conventional and/or group treatments. Self-help interventions can make a significant contribution in reaching this population. The telephone provides a unique low-cost delivery system that can expand the reach of a self-help cessation program to underserved groups of tobacco users. The primary objective is to evaluate the effectiveness of telephone-based counseling in promoting smokeless tobacco cessation among Minnesota residents. It is hypothesized that a greater proportion of individuals assigned to the telephone calling group will quit their use of smokeless tobacco products and all tobacco products compared to the comparison group not receiving calls. We plan to recruit 400 smokeless tobacco users who are interested in quitting their use of smokeless tobacco and randomize them to telephone counseling for smokeless tobacco cessation or to a comparison group that receives the same mailed self-help materials. All subjects will be assessed pre-intervention, and at 3- and 6-months.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older. Use snuff or chewing tobacco weekly. Snuff or chewing tobacco are primary tobacco use.

Exclusion Criteria:

No access to a telephone. Primary tobacco use is cigarettes, cigar or pipe tobacco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Point prevalent abstinence from all tobacco after 3 months.
  Point prevalent abstinence from all tobacco after 3 months.
Prolonged abstinence from all tobacco after 3 months.
  Prolonged abstinence from all tobacco after 3 months
Number of subjects who abstained for at least 24 hours.
  Number of subjects who abstained for at least 24 hours.

SECONDARY OUTCOMES:
Assess the relative costs of delivering the 2 interventions.
  Assess the relative costs of delivering the 2 interventions.
Use baseline data to predict successful tobacco cessation.
  Use baseline data to predict successful tobacco cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Sherwood, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States

REFERENCES:
- [Background] Boyle RG, Pronk NP, Enstad CJ. A randomized trial of telephone counseling with adult moist snuff users. Am J Health Behav. 2004 Jul-Aug;28(4):347-51. doi: 10.5993/ajhb.28.4.6. PMID 15228971